CLINICAL TRIAL: NCT01076452
Title: CSP #468 Phase II - A Comparison of Best Medical Therapy and Deep Brain Stimulation of Subthalamic Nucleus and Globus Pallidus for the Treatment of Parkinson's Disease, Phase II
Brief Title: Phase II Subthalamic Nucleus (STN) vs. Globus Pallidus (GPi) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medtronic (Industry)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 468 Phase II; VA-NINDS-01 (Other: NIH-NINDS)
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; levo-dopa; tremor; dyskinesia; subthalamic nucleus; globus pallidus
MeSH Terms: conditions — Parkinson Disease; Tremor; Dyskinesias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STN (Active Comparator): Participants were randomized to receive deep brain stimulation on STN (Subthalamic Nucleus) target.
  Interventions: Device: Bilateral Deep Brain Stimulation
- GPi (Active Comparator): Participants were randomized to receive deep brain stimulation on GPi (Globus Pallidus) target.
  Interventions: Device: Bilateral Deep Brain Stimulation

INTERVENTIONS:
Device: Bilateral Deep Brain Stimulation — The DBS site (STN or GPi) was assigned on a random basis at the time the patient enters the surgical phase of the trial.

SUMMARY:
The goal of the second phase of the study is to determine if simultaneous bilateral subthalamic nucleus stimulation or simultaneous bilateral globus pallidus stimulation is more effective in reducing symptoms of Parkinson's Disease.

DETAILED DESCRIPTION:
Deep Brain Stimulation (DBS) is a promising therapy for Parkinson's disease (PD) Whether DBS is superior to comprehensive best medical therapy or whether some patients or symptoms respond better to DBS in one area of the brain or the other is currently not known. The goals of this project are to compare the effectiveness of DBS and comprehensive medical therapy as treatments for PD (Phase I) and to compare bilateral DBS at 2 areas of the brain-the subthalamic nucleus (STN) and the globus pallidus (GPi) -to determine the most effective brain site for surgical intervention (Phase II) In this prospective, randomized, multi-center trial, 316 patients will be enrolled at 13 centers over four and a half years. Patients will initially be randomized to immediate surgery (DBS) or to 6 months of "best medical therapy". BMT arm patients will then be randomized to proceed into the DBS surgical phase of the trial. The DBS site (STN pr GPi) will be assigned on a random basis at the time the patient enters the surgical phase of the trial. Patients will be followed for two years post surgery (24 months for DBS only patients and 30 months for BMT-DBS patients) Effective 8/5/05 randomization to the BMT arm has been discontinued since the study has sufficient information to compare the outcomes of DBS and BMT patients at 6 months. The findings will be critically important in establishing the optimal surgical treatment of the disabling symptoms of PD.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's Disease
* Hoehn and Yahr stage 2 or worse when off medications
* L-dopa responsive with clearly defined "on" periods (i.e. symptoms improve at least partially with L-dopa administration, a characteristic that helps distinguish idiopathic PD from "Parkinson's Plus" and atypical Parkinson's syndromes-see below)
* persistent disabling symptoms (e.g. on troubling dyskinesias, or disabling "off" periods at least 3 hours/day) despite medication therapy. Patients will have been treated with variable doses of levodopa and dopamine agonists (at a minimum) and will have had an adequate trial of other adjunctive medications)
* stable on medical therapy for at least one month prior to study enrollment
* age >21
* available and willing to be followed-up according to study protocol

Exclusion Criteria:

* "Parkinson's plus" syndromes, secondary, or atypical Parkinson's syndromes (e.g. progressive supranuclear palsy, striato-nigral degeneration, multiple system atrophy, post-stroke, post-traumatic, or post-encephalitic Parkinson's. These patients have cardinal symptoms characteristic of PD but with additional symptoms indicating other organic brain dysfunction, such as gaze palsies, autonomic dysfunction, lack of response to L-dopa, these individuals tend not to improve with standard treatments for PD)
* previous Parkinson's Disease surgery
* medical contraindications to surgery or stimulation (e.g. uncontrolled hypertension, advanced coronary artery disease, other implanted stimulation or electronically-controlled devices including cardiac demand pacemaker, aneurysm clips, cochlear implants, or a spinal cord stimulator) (Note: for the subject who receives either a pacemaker and/or defibrillator after this study enrollment, he/she will be allowed to continue the study if the neurostimulator system can be adequately programmed to permit system compatibility)
* contraindication to magnetic resonance imaging (e.g. indwelling metal fragments or implants that might be affected by MRI)
* active alcohol or drug abuse
* score on Mini-Mental Status examination of 24 or lower, or other neuropsychological dysfunction 9e.g. dementia) that would contraindicate surgery
* intracranial abnormalities that would contraindicate surgery (e.g. stroke, tumor, vascular abnormality affecting the target area)
* pregnancy
* concurrent participation in another research protocol

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2002-04; Primary Completion 2008-10 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Follett, Study Chair — VA Medical Center, Iowa City
Locations (14):
- United States (14):
  - University of California at Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - VA Medical Center, Portland, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Philadelphia, OPC, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Medical College of Virginia, Richmond, Virginia
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Result] Weaver FM, Follett K, Stern M, Hur K, Harris C, Marks WJ Jr, Rothlind J, Sagher O, Reda D, Moy CS, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein J, Stoner G, Heemskerk J, Huang GD; CSP 468 Study Group. Bilateral deep brain stimulation vs best medical therapy for patients with advanced Parkinson disease: a randomized controlled trial. JAMA. 2009 Jan 7;301(1):63-73. doi: 10.1001/jama.2008.929. PMID 19126811
- [Result] Follett KA, Weaver FM, Stern M, Hur K, Harris CL, Luo P, Marks WJ Jr, Rothlind J, Sagher O, Moy C, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein JM, Stoner G, Starr PA, Simpson R, Baltuch G, De Salles A, Huang GD, Reda DJ; CSP 468 Study Group. Pallidal versus subthalamic deep-brain stimulation for Parkinson's disease. N Engl J Med. 2010 Jun 3;362(22):2077-91. doi: 10.1056/NEJMoa0907083. PMID 20519680
- [Result] Weaver FM, Follett KA, Stern M, Luo P, Harris CL, Hur K, Marks WJ Jr, Rothlind J, Sagher O, Moy C, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein JM, Stoner G, Starr PA, Simpson R, Baltuch G, De Salles A, Huang GD, Reda DJ; CSP 468 Study Group. Randomized trial of deep brain stimulation for Parkinson disease: thirty-six-month outcomes. Neurology. 2012 Jul 3;79(1):55-65. doi: 10.1212/WNL.0b013e31825dcdc1. Epub 2012 Jun 20. PMID 22722632
- [Result] Weintraub D, Duda JE, Carlson K, Luo P, Sagher O, Stern M, Follett KA, Reda D, Weaver FM; CSP 468 Study Group. Suicide ideation and behaviours after STN and GPi DBS surgery for Parkinson's disease: results from a randomised, controlled trial. J Neurol Neurosurg Psychiatry. 2013 Oct;84(10):1113-8. doi: 10.1136/jnnp-2012-304396. Epub 2013 May 10. PMID 23667214
- [Derived] Ostrem JL, Luo P, Weaver FM, Follett K, Rothlind J, Galifianakis NB, Lai EC, Bronstein J, Duda J, Holloway K, Sarwar A, Brodsky M, Chung K, Spindler M, Reda D, Snodgrass A, Moy C, Huang G, Wei Y, Marks WJ Jr; CSP 468F Study Group. 10-year clinical outcomes of subthalamic nucleus versus pallidal deep brain stimulation for Parkinson's disease: VA/NINDS CSP #468F. Front Neurol. 2026 Jan 16;16:1728999. doi: 10.3389/fneur.2025.1728999. eCollection 2025. PMID 41626017
- [Derived] Rothlind JC, York MK, Carlson K, Luo P, Marks WJ Jr, Weaver FM, Stern M, Follett K, Reda D; CSP-468 Study Group. Neuropsychological changes following deep brain stimulation surgery for Parkinson's disease: comparisons of treatment at pallidal and subthalamic targets versus best medical therapy. J Neurol Neurosurg Psychiatry. 2015 Jun;86(6):622-9. doi: 10.1136/jnnp-2014-308119. Epub 2014 Sep 2. PMID 25185211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 299 subjects were enrolled into the study from May 2002 to September 2006 at 13 clinical sites including 7 VA Medical Centers and 6 affiliated university medical centers.
Groups:
- Arm 1: STN (Subthalamic Nucleus)
  Bilateral Deep Brain Stimulation : The DBS site (STN or GPi) will be assigned on a random basis at the time the patient enters the surgical phase of the trial.
- Arm 2: GPi (Globus Pallidus)
  Bilateral Deep Brain Stimulation : The DBS site (STN or GPi) will be assigned on a random basis at the time the patient enters the surgical phase of the trial.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 147 | 152
Completed | 123 | 138
Not Completed | 24 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 147 | 152 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 113 | 117 | 230
  >=65 years | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (8.7) | 61.8 (8.7) | 61.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 19 | 50
  Male | 116 | 133 | 249
Region of Enrollment [Number; unit: participants]
  United States | 147 | 152 | 299

OUTCOME MEASURES:

1. Secondary Outcome: The Change From Baseline in the UPDRS Scores Part I (Mentation) at 24 Months.
Description: The UPDRS has four parts (Parts I-IV) in which a total of 42 disease characteristics are assessed. Most characteristics are assessed according to their severity on a 0-4 scale (0 = normal, 4 = most substantial impairment), and some are assessed only for absence (score = 0) or presence (score = 1). Part I has four items assessing intellectual impairment, thought disorder, depression and motivation. A summary score ranging from 0 to16 is generated by adding the four items. The higher score indicates worse condition.
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- STN (Subthalamic Nucleus): STN (Subthalamic Nucleus)
  Bilateral Deep Brain Stimulation : The DBS site (STN or GPi) will be assigned on a random basis at the time the patient enters the surgical phase of the trial.
- GPi (Globus Pallidus): GPi (Globus Pallidus)
  Bilateral Deep Brain Stimulation : The DBS site (STN or GPi) will be assigned on a random basis at the time the patient enters the surgical phase of the trial.
Arm/Group | STN (Subthalamic Nucleus) | GPi (Globus Pallidus)
Number analyzed (Participants) | 147 | 152
units on a scale | 0.6 (2.2) | 0.4 (2.2)

2. Primary Outcome: The Change From Baseline in the UPDRS-III Score at 24 Months With Deep-brain Stimulation and Without Medication.
Description: The primary outcome measure for the comparison of GPi deep brain stimulation (DBS) to STN DBS is the motor function score of the Unified Parkinson's Disease Rating Scale (UPDRS Part III) measured while the patient is off medications and on stimulation at follow-up visits post surgery. UPDRS Part III has 14 items assessing motor skills including facial expression and speech, tremors, rigidity, posture, gait, and bradykinesia. Left and right sides (arms, legs, and hands) are assessed separately for seven of the functions. The motor function (UPDRS part III) assessments are done by turning on the stimulation with and without taking PD medications (on/off) at each in-person visit. A summary score ranging from 0 to 108 is generated by adding the 14 specific motor function responses. The higher score indicates the worse motor function.
Time Frame: Baseline and 24 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | STN (Subthalamic Nucleus) | GPi (Globus Pallidus)
Number analyzed (Participants) | 147 | 152
units on a scale | -12.9 [-15.4 to -10.4] | -13.1 [-15.5 to -10.8]

3. Secondary Outcome: The Change From Baseline in the UPDRS Scores Part II (Activity of Daily Living) at 24 Months.
Description: The UPDRS has four parts (Parts I-IV) in which a total of 42 disease characteristics are assessed. Most characteristics are assessed according to their severity on a 0-4 scale (0 = normal, 4 = most substantial impairment), and some are assessed only for absence (score = 0) or presence (score = 1). Part II has 13 items focusing on activities of daily living including walking, writing, dressing and speech. A summary score ranging from 0 to 52 is generated by adding the 13 items. The higher score indicates worse condition.
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STN (Subthalamic Nucleus) | GPi (Globus Pallidus)
Number analyzed (Participants) | 147 | 152
units on a scale | -2.3 (6.6) | -3.4 (6.5)

4. Secondary Outcome: The Change From Baseline in the UPDRS Scores Part IV (Complication of Therapy) at 24 Months.
Description: The UPDRS has four parts (Parts I-IV) in which a total of 42 disease characteristics are assessed. Most characteristics are assessed according to their severity on a 0-4 scale (0 = normal, 4 = most substantial impairment), and some are assessed only for absence (score = 0) or presence (score = 1). Part IV includes four categories (11 items) related to dyskinesias, clinical fluctuations of symptoms, and other complications. A summary score ranging from 0 to 23 is generated by adding the four items. The higher score indicates worse condition.
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STN (Subthalamic Nucleus) | GPi (Globus Pallidus)
Number analyzed (Participants) | 147 | 152
units on a scale | -3.9 (3.4) | -3.4 (3.8)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events were identified rigorously and categorized as mild, moderate, or severe. Serious adverse events included any event that resulted in death, disability, prolonged or new hospitalization; was life-threatening; or required medical or surgical intervention to prevent one of the above outcomes.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 83/147 | 77/152
Other Adverse Events (participants affected / at risk) | 145/147 | 150/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=147) | Arm 2 (N=152)
Implantation-site infection (Infections and infestations) | 11 (14) | 12 (17)
Fall (Injury, poisoning and procedural complications) | 13 (16) | 5 (5)
Pneumonia (Infections and infestations) | 4 (4) | 8 (8)
Confusional state (Psychiatric disorders) | 5 (5) | 2 (2)
Medical device complication (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Lumbar spine stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Mental Status Change (Psychiatric disorders) | 1 (2) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Syncope (Nervous system disorders) | 4 (4) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 4 (4)
Adverse Drug Reaction (General disorders) | 2 (2) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 3 (3) | 1 (1)
Dyskinesia (Nervous system disorders) | 3 (3) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Suicidal Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Cerebral hemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Stroke (Nervous system disorders) | 3 (3) | 0 (0)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 2 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (2)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 1 (1)
drug hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Road Traffic accidents (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Restenosis (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis Perforated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Instestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 1 (1)
Implant Site Reaction (General disorders) | 0 (0) | 1 (1)
Mechanical Complication of Implant (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Clostridium Difficile Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Localized Infection (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=147) | Arm 2 (N=152)
Fall (Injury, poisoning and procedural complications) | 103 (198) | 100 (157)
Freezing Phenomenon (Nervous system disorders) | 65 (93) | 80 (113)
Aneamia (Blood and lymphatic system disorders) | 7 (7) | 9 (14)
Diplopia (Eye disorders) | 7 (7) | 3 (3)
Visual Disturbance (Eye disorders) | 7 (7) | 12 (12)
Constipation (Gastrointestinal disorders) | 48 (58) | 56 (65)
Dysphagia (Gastrointestinal disorders) | 66 (84) | 71 (85)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (15) | 10 (10)
Nausea (Gastrointestinal disorders) | 28 (32) | 18 (19)
Vomiting (Gastrointestinal disorders) | 6 (6) | 8 (8)
adverse drug reaction (General disorders) | 10 (12) | 7 (14)
Asthenia (General disorders) | 11 (13) | 5 (5)
Chest Pain (General disorders) | 11 (12) | 10 (10)
Fatigue (General disorders) | 26 (29) | 24 (31)
Gait Disturbance (General disorders) | 71 (94) | 70 (98)
Oedema Peripheral (General disorders) | 17 (18) | 13 (13)
Pain (General disorders) | 50 (75) | 43 (65)
Implant sight infection (Infections and infestations) | 12 (15) | 13 (19)
Pneumonia (Infections and infestations) | 7 (8) | 12 (12)
Urinary Tract Infection (Infections and infestations) | 22 (28) | 16 (29)
Incision Site Pain (Injury, poisoning and procedural complications) | 31 (33) | 30 (31)
Procedural Pain (Injury, poisoning and procedural complications) | 22 (32) | 29 (41)
Blood Pressure increase (Investigations) | 10 (12) | 10 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (26) | 9 (10)
Back Pain (Musculoskeletal and connective tissue disorders) | 22 (22) | 24 (25)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 50 (74) | 41 (61)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 (16) | 6 (8)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 15 (15)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 55 (78) | 48 (79)
Akinesia (Nervous system disorders) | 30 (41) | 33 (49)
Balance disorder (Nervous system disorders) | 63 (81) | 66 (86)
Bradykinesia (Nervous system disorders) | 47 (69) | 57 (86)
Drooling (Nervous system disorders) | 56 (68) | 51 (54)
Dyskinesia (Nervous system disorders) | 76 (116) | 62 (86)
Dystonia (Nervous system disorders) | 60 (85) | 68 (89)
Headache (Nervous system disorders) | 61 (72) | 61 (71)
memory Impairment (Nervous system disorders) | 13 (14) | 23 (24)
Motor Dysfunction (Nervous system disorders) | 52 (70) | 57 (84)
Poor Quality Sleep (Nervous system disorders) | 9 (11) | 11 (12)
Somnolence (Nervous system disorders) | 18 (19) | 18 (20)
Speech Disorder (Nervous system disorders) | 78 (105) | 70 (88)
Tremor (Nervous system disorders) | 58 (83) | 54 (79)
Abnormal Dreams (Psychiatric disorders) | 13 (14) | 13 (14)
Alcohol Abuse (Psychiatric disorders) | 10 (10) | 14 (15)
Anxiety (Psychiatric disorders) | 30 (34) | 23 (27)
Confusional State (Psychiatric disorders) | 69 (98) | 58 (79)
Depression (Psychiatric disorders) | 80 (101) | 69 (94)
Hallucination (Psychiatric disorders) | 21 (25) | 21 (26)
Insomnia (Psychiatric disorders) | 40 (47) | 35 (40)
Sexual Dysfunction (Reproductive system and breast disorders) | 13 (14) | 23 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 13 (14)
Dyspnonea (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 18 (18)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 28 (37) | 31 (44)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 12 (13)
Hypertension (Vascular disorders) | 17 (18) | 22 (28)
Orthostatic Hypotension (Vascular disorders) | 44 (66) | 42 (58)

LIMITATIONS AND CAVEATS:
We observed differences between STN and GPi DBS groups on several secondary measures but these findings should be interpreted cautiously. We did not adjust for repeated significance tests and the differences may have limited clinical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days